CLINICAL TRIAL: NCT07238998
Title: Evaluating the Clinical Effectiveness of a Motivational Interviewing-Based Conversational Mobile Application for High-Risk Drinkers
Brief Title: Clinical Effectiveness of a Motivational Interviewing-Based Conversational Mobile Application for High-Risk Drinkers
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Collaborators: BlueSignum Corporation (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 4-2025-1168
Record Dates: First submitted 2025-11-16; First posted 2025-11-20 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Alcohol Drinking; High-Risk Drinking Patterns
MeSH Terms: conditions — Alcohol Drinking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chatbot Intervention Group (Experimental): Participants assigned to the experimental arm will use a motivational interviewing-based conversational agent (chatbot) mobile application for 4 weeks beginning on the baseline assessment day (Week 0). Reassessments will occur at Week 4, marking the end of the intervention period, and at Week 16, the three-month follow-up. All efficacy analyses comparing the two groups will be conducted over the Week 0-16 evaluation period.
  Interventions: Behavioral: Motivational Interviewing-Based Conversational Agent (Mobile Chatbot)
- Waitlist Control Group (Active Comparator): Participants assigned to the waitlist control arm will not receive any intervention during the primary evaluation period (Week 0-16). They will undergo the same reassessments as the intervention group at Week 4 and Week 16. After completing the Week 16 follow-up, participants in the control arm will be offered the same 4-week chatbot intervention for ethical considerations, followed by a final assessment at Week 20. However, this post-Week-16 intervention is not included in the primary efficacy analysis.
  Interventions: Other: No Intervention (Waitlist Control)

INTERVENTIONS:
Behavioral: Motivational Interviewing-Based Conversational Agent (Mobile Chatbot) — Participants in the experimental arm will use a motivational interviewing-based conversational agent (mobile chatbot) for 4 weeks starting on the baseline assessment day (Week 0). The intervention provides daily interactive dialogues, personalized feedback, goal-setting guidance, and behavior change strategies based on motivational interviewing principles. Participants are encouraged to complete daily sessions designed to enhance motivation, support self-monitoring, and reduce high-risk alcohol consumption.
  Other Names: MI Chatbot, Digital Behavioral Intervention
  Arms: Chatbot Intervention Group
Other: No Intervention (Waitlist Control) — Participants in the waitlist control arm will not receive any intervention during the primary evaluation period (Week 0-16). They will complete the same reassessments as the intervention group at Week 4 and Week 16. After the Week 16 follow-up, control arm participants will be offered the same 4-week chatbot intervention for ethical considerations, followed by a final assessment at Week 20. This post-Week-16 intervention is not included in the primary efficacy analysis.
  Other Names: Waitlist Control, Delayed Intervention Control
  Arms: Waitlist Control Group

SUMMARY:
This study aims to evaluate and compare the degree of alcohol reduction between high-risk drinkers who use a motivational interviewing-based conversational agent (chatbot) application for four weeks and those in the control group who do not use the application, in order to verify its clinical effectiveness.

DETAILED DESCRIPTION:
"This study is a randomized controlled trial (RCT) employing a waitlist control design to examine the effectiveness of a motivational interviewing-based conversational mobile application for high-risk drinkers.

After obtaining voluntary written consent, participants will complete a screening process that includes a clinical interview (MINI, DSM) and demographic data collection. Those who meet all inclusion criteria and none of the exclusion criteria will be randomly assigned in a 1:1 ratio to either the intervention group (n = 110) or the control group (n = 110).

For the intervention group, the total study period is 16 weeks and consists of three visits (week 0, 4, and 16). The control group will participate for 20 weeks and complete four visits (week 0, 4, 16, and 20). The final follow-up assessment for both groups will be conducted via telephone and online.

The intervention group will use the mobile app (chatbot) for 4 weeks beginning on the baseline assessment day (Visit 1). Re-assessments will be conducted at week 4 (Visit 2), marking the end of the intervention period, and again at week 16 (Visit 3), which occurs three months after the intervention.

The control group will not receive any intervention from baseline to week 16 and will complete the same reassessments at week 4 (Visit 2) and week 16 (Visit 3). After the week 16 assessment, the control group will also use the mobile app for 4 weeks and undergo a final evaluation at week 20 (Visit 4), following completion of their intervention period.

This waitlist control design allows for a rigorous comparison of outcomes between the two groups while ensuring that all participants eventually receive access to the intervention, supporting both ethical considerations and improved retention.

ELIGIBILITY:
Inclusion Criteria:

1. Individuals aged 19 to 59 years who are capable of providing valid written informed consent.
2. Individuals who meet the definition of high-risk drinking (AUDIT score ≥ 8).3.- Individuals who express a desire to reduce their alcohol consumption.
3. Individuals who own and use an Android smartphone (version 8 or higher).
4. Individuals who have no difficulty using mobile applications.
5. Individuals who are able to communicate adequately with the research team.
6. Individuals who fully understand the study procedures and voluntarily agree to participate.

Exclusion Criteria:

1. Individuals who are unable to read or understand the consent form (e.g., illiterate individuals, non-Korean speakers).
2. Individuals with impaired decision-making capacity.
3. Pregnant individuals or those planning to become pregnant during the study period.
4. Individuals who are currently participating in another clinical study.
5. Individuals who are receiving treatment or counseling for alcohol-related problems.
6. Individuals who use two or more mobile phones.
7. Individuals who are expected to change their mobile phone or SIM card, or who plan to travel 8. abroad during the intervention period.
8. Any individual deemed inappropriate for study participation at the discretion of the investigator.

Ages: 19 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 220 (Estimated)
Dates: Start 2025-12-19 (Estimated); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Change in Past 7-Day Alcohol Consumption (Standard Drinks and Binge Drinking Frequency) From Baseline to Week 16 | Week 0 (Baseline), Week 4, and Week 16
  Alcohol consumption during the past 7 days-including total standard drink units and binge drinking frequency-will be assessed at Week 0, Week 4, and Week 16 using validated self-report measures. The primary efficacy analysis will evaluate changes from baseline to Week 16 in both past 7-day standard alcohol consumption and past 7-day binge drinking episodes to determine the intervention's effectiveness in reducing high-risk alcohol use.

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided